CLINICAL TRIAL: NCT05166837
Title: A Randomized, Double-blind, Placebo-controlled, Single-ascending Dose Phase Ⅰa Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of STSA-1002Following Intravenous Infusion in Healthy Subjects
Brief Title: The Safety of STSA-1002 Following Intravenous Infusion in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSA-1002-02
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1:2mg/kg (Experimental): All participants (fasted) received either 2 mg/kg of STSA-1002 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1002 injection; Drug: Placebo
- Cohort 2:5mg/kg (Experimental): All participants (fasted) received either 5 mg/kg of STSA-1002 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1002 injection; Drug: Placebo
- Cohort 3:10mg/kg (Experimental): All participants (fasted) received either 10 mg/kg of STSA-1002 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1002 injection; Drug: Placebo
- Cohort 4:20mg/kg (Experimental): All participants (fasted) received either 20 mg/kg of STSA-1002 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1002 injection; Drug: Placebo
- Cohort 5:30mg/kg (Experimental): All participants (fasted) received either 30 mg/kg of STSA-1002 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1002 injection; Drug: Placebo

INTERVENTIONS:
Drug: STSA-1002 injection — Intravenous injection
  Arms: Cohort 1:2mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 1:2mg/kg
Drug: STSA-1002 injection — Intravenous injection
  Arms: Cohort 2:5mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 2:5mg/kg
Drug: STSA-1002 injection — Intravenous injection
  Arms: Cohort 3:10mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 3:10mg/kg
Drug: STSA-1002 injection — Intravenous injection
  Arms: Cohort 4:20mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 4:20mg/kg
Drug: STSA-1002 injection — Intravenous injection
  Arms: Cohort 5:30mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 5:30mg/kg

SUMMARY:
A randomized, double-blind, placebo-controlled, single-ascending dose Phase Ⅰa study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of STSA-1002 following intravenous infusion in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, aged ≥ 18 but ≤ 65, male and female;
* Body mass index: 18.0 -25.0 kg/m2, inclusive;
* Subjects (including their partners) agree to take highly effective contraceptive measures during the study, and they have no birth plan or sperm donation plan within 5 months after the end of the study;
* Medical histories, physical examinations, laboratory examinations and study-related examinations and tests of the subjects show normal results or mild abnormalities with no clinical significance before enrollment, and the Investigator judges that they are eligible;
* Subjects are aware of the risks of the study, and voluntarily participate in the clinical study and sign an informed consent form (ICF).

Exclusion Criteria:

* Past history of tuberculosis, history of contact with active tuberculosis, and positive tuberculin test results;
* History of cardiovascular, respiratory, kidney, liver, metabolism, endocrine, gastrointestinal, blood, nerve, skin and mental illness, cancer or other major disease that in the judgment of the Investigator might put the subject as risk on this study;
* There is a clear history of food or drug allergy or the total serum immunoglobulin IgE is higher than the upper limit of normal;
* Positive screening test results for human immunodeficiency virus (HIV-1/HIV-2) antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCVAb);
* Presence of clinically significant vital signs values or of electrocardiogram (ECG) abnormalities during the screening period, as defined by an Investigator;
* ANA positive;
* During the screening period, the white blood cell count and C-reactive protein test results are abnormal and have clinical significance, hemoglobin: male <120g/L or female <110g/L;
* Smoking more than 5 cigarettes per day or equivalent amount of tobacco in the 3 months before screening;
* Subjects whose daily consumption of alcohol at the time of screening or at any time within the prior 6 months is more than 2 standard drinks, where 1 standard drink = 355 mL or 12 oz (1 can) of regular-strength (5%) beer; 150 mL or 5 oz wine; 45 mL or 1.5 oz liquor/spirits (40%);
* Subjects who had a history of drug abuse or tested positive for drugs within 1 year before screening;
* Subjects who have donated either more than approximately 500 mL of blood (exclusive plasma donation) within 3 mooth prior to screening or any plasma within 4 weeks prior to screening;
* Participate in any drug or vaccine clinical trial as a subject within 3 months before screening or prepare to be vaccinated during the study period to 2 months after the end of the study;
* Have taken drugs that may affect immune function within 6 months before screening or have received any monoclonal antibody or biological agent treatment within the previous 3 months and have taken prescription/over-the-counter drugs, herbal medicines, vitamins or other supplements within the previous 14 days;
* Drink more than 5 cups of coffee, tea or cola per day (150ml and above per cup);
* Women who are pregnant or breastfeeding;
* People with a history of fainting, bleeding and needles;
* The investigator believes that there are any subjects who are not suitable to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Clinically Significant Laboratory Abnormalities, Clinically Significant Electrocardiogram Abnormalities, Clinically Significant Vital Signs Abnormalities And Clinically Significant Physical Examination Abnormalities. | 48 days
Maximum plasma concentration (Cmax) | Up to 1152 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Area under the plasma concentration-time curve from time 0 to the collection time point t of the last measurable concentration (AUC0-t) | Up to 1152 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-∞) | Up to 1152 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Time of maximum concentration (Tmax) | Up to 1152 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Elimination half-life (t1/2) | Up to 1152 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Elimination rate constant of plasma drug concentration in terminal phase (λz) | Up to 1152 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Last measurable concentration (Clast) | Up to 1152 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Mean residence time (MRT) | Up to 1152 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Clearance (CL) | Up to 1152 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Apparent volume of distribution (Vz) | Up to 1152 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects

SECONDARY OUTCOMES:
Change from baseline in concentration of free C5a and anti-drug antibody | Up to 1152 hours postdose
  To evaluate the pharmacodynamics (PD) characteristics and immunogenicity of STSA-1002 in healthy subjects
Change from baseline in concentration of CH50, IL-6, IL-8,C4, TNF-α, IFN-γ | Up to 1152 hours postdose
  To evaluate the effect of STSA-1002 on CH50, IL-6, IL-8, C4,TNF-α, IFN-γ

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The second hospital of Anhui medical university, Hefei, Anhui
  - Peking university People's Hospital, Beijing, Beijing Municipality
  - The fifth affiliated hosipital of Guangzhou medical university, Guangzhou, Guangdong
  - Peking university Shenzhen Hospital, Shenzhen, Guangdong
  - The affiliated hospital of Guizhou medical university, Guiyang, Guizhou

IPD SHARING:
Plan to Share IPD: No